CLINICAL TRIAL: NCT07394218
Title: Study on ctDNA-guided Treatment Decision-making for HER2-negative Metastatic Breast Cancer
Brief Title: ctDNA-guided Treatment Decision-making
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Prof. Hongxia Wang, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECISION
Record Dates: First submitted 2025-12-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer ( HER2 Negative); ctDNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADC + Ivonescimab (Experimental): Patients with <50% mean ctDNA VAF reduction receive ADC combined with ivonescimab.
  Interventions: Drug: ADC; Drug: Ivonescimab
- ADC Monotherapy (Active Comparator): Patients with <50% mean ctDNA VAF reduction receive continued ADC monotherapy.
  Interventions: Drug: ADC
- ADC Monotherapy (ctDNA responder cohort) (Active Comparator): Patients with ≥50% mean ctDNA VAF reduction continue ADC monotherapy.
  Interventions: Drug: ADC

INTERVENTIONS:
Drug: ADC — ADC therapy includes sacituzumab govitecan or trastuzumab deruxtecan administered intravenously according to standard dosing schedules. ADC treatment is given in all study stages and continued until disease progression or unacceptable toxicity.
Drug: Ivonescimab — Ivonescimab is administered intravenously at 20 mg/kg every 3 weeks in combination with ADC therapy for patients assigned to the combination treatment arm.
  Arms: ADC + Ivonescimab

SUMMARY:
This is an exploratory, ctDNA-guided, multi-stage clinical study designed to evaluate the clinical value of treatment decision-making based on circulating tumor DNA (ctDNA) variant allele frequency (VAF) dynamics in patients with HER2-negative metastatic breast cancer.

All enrolled patients will receive antibody-drug conjugate (ADC) therapy for two cycles in Stage 1, with serial ctDNA assessments performed prior to Cycle 1 and Cycle 2. In Stage 2, patients without disease progression will be assigned to different treatment strategies based on the percentage reduction in mean ctDNA VAF.

The study aims to assess whether ctDNA VAF dynamics can serve as an early biomarker to guide treatment intensification and improve clinical outcomes in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years；ECOG performance status 0-1； Histologically or cytologically confirmed HER2-negative metastatic breast cancer； At least one measurable lesion per RECIST v1.1； Eligible for ADC therapy； Adequate organ and bone marrow function； Life expectancy ≥3 months； Willingness to provide tumor tissue and blood samples； Signed informed consent

Exclusion Criteria:

* Prior treatment with ADC targeting the same antigen and payload；History of grade ≥3 immune-related adverse events； Active or untreated CNS metastases； Active autoimmune disease requiring systemic therapy； Clinically significant cardiovascular disease； Active interstitial lung disease； Active infection including tuberculosis, HIV, hepatitis B or C； Pregnancy or breastfeeding；Investigator-determined conditions that may interfere with study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in TNBC (Group A vs Group B) | From randomization until progression or death (up to 36 months)
  Time from randomization to disease progression or death, assessed by RECIST v1.1.

SECONDARY OUTCOMES:
ORR (RECIST v1.1)，DoR，CBR，OS，Safety (CTCAE v5.0) | From treatment initiation until end of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No